CLINICAL TRIAL: NCT03305744
Title: Atrial Electromechanical Function in Middle-aged Endurance Athletes With and Without Atrial Fibrillation
Brief Title: Atrial Electromechanical Function in Endurance Athletes With and Without Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Emily Vecchiarelli, Principal Investigator, University of Toronto
Other Study IDs: AthletesHeartUofT
Record Dates: First submitted 2017-09-29; First posted 2017-10-10 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Athlete; Middle-aged; Endurance training; Cardiac Function; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endurance Athlete with Atrial Fibrillation: These are middle-aged athletes who are diagnosed with paroxysmal Atrial Fibrillation in the last 4 years, but are otherwise free of disease.
- Endurance Athlete without Atrial Fibrillation: These are middle-aged athletes who will serve as our control group- they have not been diagnosed with AF or any other disease.

SUMMARY:
This study evaluates cardiac structure and function differences between healthy endurance trained athletes with atrial fibrillation and healthy age matched endurance trained athletes without atrial fibrillation. It is hypothesized that despite having similar structural adaptations of the heart (due to endurance training), athletes with atrial fibrillation display will impaired heart functional measures compared to endurance athletes without atrial fibrillation.

DETAILED DESCRIPTION:
Regular physical activity, including vigorous exercise, lowers cardiovascular risk factors, including the risk of developing Atrial Fibrillation (AF), one of the most commonly diagnosed types of arrhythmias. Paradoxically, despite the cardioprotective effects of exercise, middle aged endurance athletes are at 5 fold risk of developing AF compared to active individuals. Long standing endurance training induces significant changes to the heart- collectively known as the 'athlete's heart.' While these changes may be beneficial for performance, they may be conducive in promoting the risk of AF in this cohort. The aim of this study is to compare cardiac structure and function in endurance athletes diagnosed with AF (n=17) and in healthy aged matched endurance athletes (n=17). Male subjects between ages 45 and 65 years old with a long-standing history of endurance training and competition will be recruited. Heart structure and function will be compared at rest and during submaximal exercise. Participants will also complete fitness assessments and questionnaires that characterize their lifetime involvement in exercise training. This study will address the gap in the literature regarding the interaction of endurance training and AF risk.

ELIGIBILITY:
Inclusion Criteria:

ALL participants:

* endurance athlete (cyclist, runner, triathlete or other) who participate in vigorous year-round training of 4-6 hours per week for a minimum of 20 years
* participation in atleast one major competition per year (marathon/triathlon/endurance competition)
* sinus rhythm during all assessments

Inclusion criteria specific to endurance athletes with AF:

* diagnosed with lone paroxysmal AF in the last 4 years
* able to verify diagnosis (ECG or Holter verification/proof of diagnosis),
* can be on any type of medication.

Inclusion criteria specific to healthy endurance athletes without AF:

* previous participation in Athlete's Heart Study
* has completed resting cardiac magnetic resonance imaging and resting electrocardiogram

Exclusion Criteria:

* females
* no more than >1 hour per week of resistance training
* treatment or prior diagnosis of cardiovascular disease, valvular disease, hypertension, heart failure, diabetes, thyroid disorder, sleep apnea, current/recent viral disease, chronic inflammatory disease
* previous (within 10 years) or current smoking
* recreational drug use or alcohol consumption in excess of accepted standards
* inability to provide informed consent
* inability to verify AF diagnosis (if AF athlete).

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample from, but not limited to, various running, cycling, and rowing clubs for middle-aged athletes. Healthy endurance athletes will be selected from an existing study for convenience (non-probability sample). Endurance athletes with AF will be selected from the community (probability sample).
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Left intra-atrial electromechanical delay (ms) | baseline (day 1: at first visit, one time measure)
  Left intra-atrial electromechanical delay will be measured using cardiac echocardiography at rest and during submaximal cycling. Left intra-atrial electromechanical delay will be measured as the time interval between the initiation of the P wave (on an electrocardiogram) to the beginning of the late diastolic wave (Am wave) on echocardiography.

SECONDARY OUTCOMES:
Left atrial reservoir function | baseline (day 1: at first visit, one time measure)
  Left atrial reservoir function will be measured by Speckle Tracking echocardiography, at 60-80 frames per second. Left atrial reservoir function will be measured by assessing left atrial reservoir strain (%), measured during ventricular systole on echocardiography.
Left atrial volume (mL) | baseline (day 1: at first visit, one time measure)
  Left atrial volume (mL) will be measured using echocardiography at the end of ventricular systole, prior to the opening of the mitral valve. Imaging will be acquired using two and four chamber views.

OTHER OUTCOMES:
Lifetime hours of Physical Activity (# of hours) | baseline (day 1: at first visit, one time measure)
  Total lifetime hours of physical activity will be assessed using the Lifetime Physical Activity Questionnaire (LTPAQ).
Maximal oxygen consumption (VO2 max) | baseline (day 1: at first visit, one time measure)
  Maximal oxygen consumption (VO2 max) will be determined using a maximal treadmill test, in which a calibrated metabolic cart and indirect calorimetry will be used. VO2 max will be expressed as ml/kg/min.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Vecchiarelli, BKin, Principal Investigator — University of Toronto; Jack Goodman, PhD, Principal Investigator — University of Toronto; Paul Dorian, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- Goldring Center for High Performance, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Participant data may be used for future study upon participant consent for their de-identified data to be used in the event that a related study is conducted. Only principal investigators will have access to records and will have the ability to share data with approved researchers.

REFERENCES:
- [Background] Molina L, Mont L, Marrugat J, Berruezo A, Brugada J, Bruguera J, Rebato C, Elosua R. Long-term endurance sport practice increases the incidence of lone atrial fibrillation in men: a follow-up study. Europace. 2008 May;10(5):618-23. doi: 10.1093/europace/eun071. Epub 2008 Apr 4. PMID 18390875
- [Background] Grimsmo J, Grundvold I, Maehlum S, Arnesen H. High prevalence of atrial fibrillation in long-term endurance cross-country skiers: echocardiographic findings and possible predictors--a 28-30 years follow-up study. Eur J Cardiovasc Prev Rehabil. 2010 Feb;17(1):100-5. doi: 10.1097/HJR.0b013e32833226be. PMID 20065854
- [Background] Calvo N, Brugada J, Sitges M, Mont L. Atrial fibrillation and atrial flutter in athletes. Br J Sports Med. 2012 Nov;46 Suppl 1:i37-43. doi: 10.1136/bjsports-2012-091171. PMID 23097477

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT03305744/Prot_SAP_000.pdf